CLINICAL TRIAL: NCT04257994
Title: Analysis of Distribution of Cell-cell Junction Proteins in Buccal Smear Samples From Patients With Arrhythmic Disorders and Family Members at Risk as a Means for Diagnosis
Brief Title: Distribution of Cell-cell Junction Proteins in Arrhythmic Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: St. George's Hospital, London (Other)
Responsible Party: Principal Investigator, ANGELIKI ASIMAKI, Senio Lecturer in Cardiac Morphology and Sudden Death, St. George's Hospital, London
Other Study IDs: 16.0099
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Arrhythmogenic Right Ventricular Dysplasia; Brugada Syndrome; Cardiac Channelopathy
Keywords: cardiac arrhythmias
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Brugada Syndrome; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with arrhythmic disorders: Participants will include patients diagnosed with a heritable arrhythmic disorder (including arrhythmogenic, hypertrophic and dilated cardiomyopathy, cardiac sarcoidosis as well as cardiac channelopathies; Long QT syndrome, Brugada syndrome and catecholaminergic polymorphic ventricular tachycardia) followed at the Inherited Cardiac Conditions (ICC) service of St. George's University Hospitals NHS Foundation Trust as well as family members of victims of SCD evaluated at the same clinic for risk assessment and diagnosis.
  Interventions: Diagnostic Test: obtaining a buccal smear sample

INTERVENTIONS:
Diagnostic Test: obtaining a buccal smear sample — A sample will be taken from the inside of the participants' cheeks using a soft brush

SUMMARY:
Every week in the UK, 12 apparently healthy and fit individuals under the age of 35 die suddenly, a tragic event known as sudden cardiac death (SCD). The investigators have shown that heritable cardiac disorders affect the distribution of proteins at the cardiac cell-cell junctions, the areas where cardiac cells are mechanically and electrically coupled. This knowledge has helped the investigators diagnose specific heart disorders in individuals thus reducing the risk and incidence of SCD. Yet, the primary material required is a heart sample. A heart biopsy is an invasive process that comes with risks and is not performed unless absolutely necessary. And it is impossible to obtain a heart sample from an individual that may be carrying a disease-causing mutation (and hence be at risk of SCD) but does not yet show evidence of disease manifestation. The investigators recently showed that buccal cells show changes in protein distribution equivalent to those exhibited by the heart,hence providing them with a surrogate tissue for the myocardium. The investigators aim to use buccal smears as a means to identify those at risk of SCD. Patients regularly seen at the cardiology clinics at St. George's Hospital can participate in the study. The investigators shall take a buccal smear simply by rubbing a soft brush at the inside of their cheek and smearing it on a slide. Most individuals willing to participate in the study will only have to provide the investigators with a sample once. However, in selected cases (for instance, if the patients show disease progression or have a change in medication) they may be asked to provide the investigators with a subsequent sample during one of their scheduled follow-up visits. The process takes only a few seconds, is totally risk- and pain-free and it is anticipated to have great implications in diagnosis and patient management.

DETAILED DESCRIPTION:
Exfoliated buccal mucosa cells have been used as a source of material for various genetic tests and in studies of oral cancer but their use in studies of cardiovascular disease has been limited. Previous applications have included analysis of telomere length in buccal cells from patients with ischemic heart failure and measurements of intracellular magnesium levels in patients undergoing radiofrequency catheter ablation for atrial fibrillation. To the best of the investigators' knowledge, their study published at Circulation Arrhythmia and Electrophysiology 9(2) in 2016, was the first analysis of buccal mucosa cells in patients with a heritable form of heart disease. This analysis included 39 patients diagnosed with arrhythmogenic cardiomyopathy (ACM), a primary myocardial disease characterized by an unusually high burden of arrhythmias and sudden cardiac death as well as 15 carriers of disease-causing mutations without overt disease manifestation. In a subsequent analysis (unpublished data), 55 additional individuals affected by ACM were sampled and the positive predictive value of our approach in diagnosing the disease was 91.9%. Although highly arrhythmogenic, ACM is a relatively rare disorder. The investigators are now at a position to apply this simple, totally risk-free approach to help identify those individuals at risk of SCD due to more common forms of heritable arrhythmic disorders including the cardiac channelopathies. The cardiologists at St. George's University of London evaluate more than 100 families of SCD victims per year for diagnosis and risk assessment. The large number of individuals evaluated at this single site provides the unprecedented opportunity to use this novel diagnostic approach to aid significant numbers of those at risk of developing life-threatening arrhythmias. There are no risks or potential discomfort associated with the study for the volunteer participants. The outcomes, however, may prove highly beneficial for prevention of SCD, timely and accurate diagnosis and management of arrhythmic disorders.

The study participants will just be asked to open their mouth. A study team member will rub a soft brush a few times at the inside of their cheek and smear the brush on a microscopy slide. The slide will be sprayed with 70% ethanol to preserve the material and taken to the research laboratory where it will be subjected to immunostaining to study the distribution of key proteins. The patient will have a total of 4 smears taken (2 from each cheek). For the majority of the patients, only a single sampling will be enough which will take place during one of their regular follow-up appointments at the cardiology clinic. There is no pain and no discomfort associated with the procedure and it lasts only a few seconds. In selected cases, however, if for instance the investigators want to use the buccal smear to evaluate the effect of a novel drug treatment on protein distribution, the patient might be asked to provide the study team with another sample, again during one of his scheduled regular follow-up visits

ELIGIBILITY:
Inclusion Criteria:• Participants will include patients diagnosed with a heritable arrhythmic disorder (including arrhythmogenic, hypertrophic and dilated cardiomyopathy, cardiac sarcoidosis as well as cardiac channelopathies; Long QT syndrome, Brugada syndrome and catecholaminergic polymorphic ventricular tachycardia) followed at the Inherited Cardiac Conditions (ICC) service of St. George's University Hospitals NHS Foundation Trust.

* Family members of victims of SCD evaluated at the same clinic for risk assessment and diagnosis. These groups include both individuals with clear disease manifestation (termed "affected") as shown by conventional diagnostic approaches (electrocardiography, echocardiography, cardiac MRI, Holter monitoring) as well as potential carriers of disease-causing mutations who, however, may not/not yet manifest any overt sign of cardiovascular abnormalities (termed "carriers"). These are typically family members of probands diagnosed with a heritable arrhythmic disorder or family members of a sudden cardiac death victim.
* All individuals that fall in the above categories will be included regardless of their management (medication, devices, and surgical procedures).
* Individuals with co-existing conditions will also be included and their medical history will be taken into account when interpreting the results of the immunohistochemical analysis.
* Adult individuals (>18 years of age).
* Pregnant women will be included as the approach used is not in any way harmful or uncomfortable.
* All individuals must have provided the study team with a signed informed consent in order to participate in the study.

Exclusion Criteria:• Children under 18 years of age

* Individuals lacking decisional capacity.
* Individuals with non-heritable, non-arrhythmic cardiac disorders (such as ischemic heart disease or inflammatory disorders) followed at St. George's University Hospitals NHS Foundation Trust.
* Non-English speakers will be excluded from the study unless a translator is present who can thoroughly explain to them the research question/plan in order for them to provide an informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will include individuals that have arrhythmic disorders or are being evaluated for arrhythmic disorders due to a family history of sudden cardiac death at the cardiology center of St George's.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2027-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Angeliki Asimaki, Principal Investigator — St George's, University of London
Locations (1):
- St George'S Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Predisposed for Heritable Cardiac Disorder: Eligible participants will either have a diagnosis of a heritable heart condition or be a relative of a sudden cardiac death victim/ person diagnosed with a heritable heart condition
Period: Overall Study
Arm/Group | Predisposed for Heritable Cardiac Disorder
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Arrhythmic Disorders
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: Alteration of Key Protein Distribution
Description: We recruit individuals that have propensity to an arrhythmic disorder (ie. they are carriers of disease-causing mutations) or they have been already diagnosed with a heritable heart condition.
  The primary outcome measure is whether key proteins show altered localization in the eligible participants.
  We are reporting the number of participants that did show altered protein distribution at baseline. There is no unit of measurement for this outcome. Cheek smears are subjected to immunofluorescence staining and examined under a confocal microscope. The technique has been optimized to show a binary outcome: a protein is either at its normal location or not.
Time Frame: This is a longitudinal study. Each participant will provide cheek smears at recruitment to assess baseline protein distribution. Thereafter, each participant will be asked to provide follow-up samples every 6 months for the duration of the study.
Population: bearing a heritable heart disease mutation or be a first degree relative of SCD victim of carrier of heart disease mutation
Measure: Count of Participants; unit: Participants
Groups:
- Predisposed for Heritable Cardiac Disorder: Eligible participants will either have a diagnosis of a heritable heart condition or by at risk of developing an arrhythmic disorder (ie. are carriers of disease-causing mutations)
Arm/Group | Predisposed for Heritable Cardiac Disorder
Number analyzed (Participants) | 26
Participants | 26

2. Secondary Outcome: Correlation of Protein Distribution With Participants' Genotype
Description: A potential secondary outcome of the research is whether the investigators can correlate protein distribution in the buccal mucosa with specific genotypes. The investigators' preliminary results on the cohort of patients with ACM suggest that mutations in different genes result in different protein distribution patterns within the buccal mucosa. Being able to predict the gene bearing the disease-causing mutation will significantly reduce the time and cost of genetic sequencing. Identifying the specific gene underlying a heritable arrhythmic disorder is of pivotal importance as increasingly developing genotype/phenotype correlations help individualized risk identification and patient management.
Time Frame: as for outcome 1
Reporting Status: Not Posted

3. Secondary Outcome: Correlation of Treatments With Cx43 Distribution
Description: Another potential outcome has to do with the effect changes in the patients' treatment plans may have on Cx43 distribution. Cx43 is the major gap junction protein responsible for the electrical coupling of the cells. It has been shown that patients with arrhythmic disorders show decreased distribution of Cx43 at the cell borders in their hearts and this has been associated with an increased risk for arrhythmias. The investigators' preliminary studies show that patients with cardiomyopathies show Cx43 remodeling in their buccal mucosa. If a patient seen at the arrhythmia service of St. George's shows Cx43 remodeling during initial sampling and in a follow-up visit his clinical care team deems necessary to change his treatment plan the investigators would like to study Cx43 distribution again during one of his/hers follow up visits. If the new treatment plan results in restoration of Cx43, this finding may be an indication of successful arrhythmia management.
Time Frame: as for outcome 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: through study completion an average of 1 year
Description: no adverse events recorded
Arm/Group | Predisposed for Heritable Cardiac Disorder
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Predisposed for Heritable Cardiac Disorder (N=18)
no adverse events recorded (Congenital, familial and genetic disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT04257994/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT04257994/ICF_001.pdf